CLINICAL TRIAL: NCT06534593
Title: Effects of Physical Therapy on Low Back Pain, Disc Height Index, Postural Stability, Disability, Gait and Function in Persons With Postero-lateral Disc Herniation: The DISC-RELIEF Trial
Brief Title: Effects of Physical Therapy on Low Back Pain, Disc Height Index, Postural Stability, Disability, Gait and Function in Persons With Postero-lateral Disc Herniation
Acronym: DISC-RELIEF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/16
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Herniation, Disc; Low Back Pain
MeSH Terms: conditions — Intervertebral Disc Displacement; Low Back Pain | interventions — Electric Stimulation Therapy; Diathermy

STUDY DESIGN:
Intervention Model Description: the study will consist of 2 arms.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The Control group will receive standard treatment for the management of discogenic low back pain.
  Interventions: Other: Standard medical treatment
- Experimental Group (Experimental): The Physical Therapy group will receive Physical Therapy for the management of discogenic low back pain.
  Interventions: Device: Lumbar Traction; Other: Mckenzie Extension Protocol; Device: Interferential Therapy; Device: Heat Therapy; Other: Sustained Natural Apophyseal Glides (SNAGs)

INTERVENTIONS:
Other: Standard medical treatment — Standard medical treatment
  Arms: Control Group
Device: Lumbar Traction — Lumbar traction using traction table
  Arms: Experimental Group
Other: Mckenzie Extension Protocol — Mckenzie Extension Exercises
  Arms: Experimental Group
Device: Interferential Therapy — Interferential Therapy for 20 minutes
  Arms: Experimental Group
Device: Heat Therapy — Heat Therapy for 20 minutes
  Arms: Experimental Group
Other: Sustained Natural Apophyseal Glides (SNAGs) — 3-5 reptations of Mulligan's lumbar extension Sustained Natural Apophyseal Glides (SNAGs)
  Arms: Experimental Group

SUMMARY:
The current study aims to determine if physical therapy is significantly superior in improving postural stability, pain and function and disc height index in persons with discogenic low back pain, as compared to the standardized medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female participants
* Postero-lateral lumbar disc herniation
* Aged 18-50 years old
* Low back pain intensity less than 80/100mm on visual analogue scale or 8/10 on numeric pain rating scale
* Positive peripheralization and centralization phenomenon

Exclusion Criteria:

* Individuals with and any musculoskeletal, metabolic, or neurological disorders that may impair gait, postural stability or sensory integrity will be excluded from the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-08-07 (Estimated); Primary Completion 2025-02-07 (Estimated); Study Completion 2025-02-07 (Estimated)

PRIMARY OUTCOMES:
Back Pain | 2 weeks
  Pain will be measured via Visual Analogue Scale. A higher score signifies poor outcome.
Lumbar Range of Motion | 2 weeks
  Lumbar Range of Motion will be measured via inclinometer. A higher score signifies good outcome.
Postural Stability | 2 weeks
  Postural Stability will be measured via Biodex Balance System. A higher score signifies poor outcome.
Lumbar Disability | 2 weeks
  Lumbar Disability will be measured via Oswestry Disability Index.
Stride length | 2 weeks
  Stride length during gait will be analyzed using observational gait analysis. A greater stride length signifies better outcome
Gait Velocity | 2 weeks
  Velocity during gait will be analyzed using observational gait analysis. A greater gait velocity signifies better outcome
Cadence | 2 weeks
  Cadence during gait will be analyzed using observational gait analysis, which is number of steps per minute.
Disc height index | 2 weeks
  Disc height index will be analyzed using Magnetic Resonance Imaging. A greater disc height index signifies better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Osama, PhD*, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation University Islamabad, Islamabad, Federal, Pakistan